CLINICAL TRIAL: NCT07326748
Title: Development and Evaluation of an Indigenized Family Acceptance Project for Lakota LGBTQ2S+ Youth
Brief Title: Lakota Family Acceptance Project
Acronym: L-FAP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Katie M Edwards, Professor, School of Social Work, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HUM00264029; 7R34MH134937-02 (NIH)
Record Dates: First submitted 2026-01-07; First posted 2026-01-08 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: LGBTQ; Racial Disparities; Family Relationships; Minority Stress; Depression; Anxiety; Drug Use; Teen Dating Violence; Sexual Risk Reduction
Keywords: family acceptance; LGBTQ; 2SLGBTQ+; youth; family support; parents of LGBTQ youth; Racial/Ethnic Minority; health equity; Native American/Indigenous; Two Spirit
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Other): There is only one arm in this OPT and that is the intervention group that will participate in the 8-session LFAP intervention
  Interventions: Behavioral: Adapted Lakota Family Acceptance Program

INTERVENTIONS:
Behavioral: Adapted Lakota Family Acceptance Program — Tiwahe Tewichaglapi ("The Family Loves Them") Program Overview
  Tiwahe Tewichaglapi is a culturally grounded, family-centered intervention adapted from the Family Acceptance Project® (FAP) to promote caregiver acceptance, respect, support, and family bonding for 2SLGBTQ+ Lakota youth. The program was developed in partnership with the Lakota Oyate to address family rejection rooted in colonization and historical trauma and to honor traditional Two Spirit roles that have long held important and respected places within Lakota communities. The program aims to strengthen families, increase youth pride and hope for the future, and reduce mental health risks such as depression, anxiety, substance use, dating violence, and suicide among 2SLGBTQ+ Lakota youth.
  Tiwahe Tewichaglapi includes eight family-centered group sessions delivered by Lakota facilitators. Each session begins with Lakota cultural and spiritual practices - including smudging, a Lakota prayer, and a shared meal - to ground the

SUMMARY:
The goal of this open pilot trial (OPT) is to develop a Lakota-adapted Family Acceptance Project (LFAP) for Indigenous 2SLGBTQ+ youth and their caregivers. The OPT is specifically focused on acceptability, feasibility, and safety of programming and research protocols. The investigators will also examine pre- to post- changes on outcomes for the sole purposes of making sure scores on measures are changing in the hypothesized direction (e.g., depression scores are going from moderate to minimal as opposed to no change or depression scores increasing). Once enrolled in the study, participants complete a baseline survey. Then participants will engage in LFAP which is an 8-session group intervention; sessions will be scheduled once a week for eight weeks (at 2 hours per session). Participants will complete survey instruments before and immediately after the program sessions, in addition to post-program surveys and an exit interview.

DETAILED DESCRIPTION:
Research shows that Indigenous Lesbian, Gay, Bisexual, Transgender, Queer, and Two-Spirit (2SLGBTQ+) youth experience high rates of mental health problems. A key factor that leads to these challenges is family rejection (family behaviors and reactions that minimize, deny, ridicule and attempt to prevent or change a child's sexual orientation, gender identity and gender expression).

Family rejection among Indigenous 2SLGBTQ+ youth is rooted in colonization and multiple historical traumas. This includes disrupting traditional childrearing practices by forced placement in boarding schools that with other historical traumas focused on erasing Indigenous culture, including positive Two Spirit histories. Indeed, in many traditional Indigenous communities, including among the Lakota Oyate, Two Spirit relatives held important and honorable roles.

The Family Acceptance Project® (FAP) is a research, education and intervention program that was founded more than 20 years ago to help ethnically, racially and spiritually/religiously diverse parents and caregivers to learn to support and advocate for their 2SLGBTQ+ children and youth to prevent health and mental health problems and promote well-being. FAP conducted the first research on sexual minority and gender diverse youth and families and developed the first family support model to decrease family rejection and increase acceptance and support. FAP's work is grounded in the family's culture and spirituality/faith traditions.

The overall goal of the Tiwahe Tewichaglapi ("the family loves them" in Lakota) program is to apply FAP's culture-based model in the context of Lakota culture, history, and virtues. The investigators are carrying out this working partnership with community leadership to provide key family support services to 2SLGBTQ+ Lakota youth and their caregivers.

The open pilot trial (OPT) is specifically focused on assessing acceptability, feasibility, and safety of programming and research. The investigators will also use surveys to help us learn if the program impacts the project's goals above. Investigators will also ask SGMY and caregivers to share what they liked about the program and their guidance for enhancing it. This data will be used to further refine L-FAP prior to the start of the pilot RCT.

The goals of the program are to:

1. Promote parent/caregiver acceptance, respect, and support for their 2SLGBTQ+ Lakota youth.
2. Increase family bonding, love, support, and communication.
3. Increase LGBTQ2S+ youths' feelings of pride and hope about the future.
4. Reduce problems such as depression, anxiety, substance abuse, dating violence, and suicide.
5. Promote bright, happy, and thriving futures for 2SLGBTQ+ Lakota youth.

Before receiving Tiwahe Tewichaglapi, SGMY (ages 13 to 18) and their caregivers will complete a survey. After completing this initial (baseline) survey, half of the families will participate in program sessions. Following the first round of sessions, all participants will complete an immediate follow-up survey. After this final survey, the other half of families will attend the program sessions.

The project includes an Advisory Board with representation from 2SLGBTQ+ Lakota youth, their caretakers, and professionals who work with 2SLGBTQ+ Lakota youth and their families, Elders and Spiritual Leaders. These individuals will provide input on key aspects of the project to ensure that it is culturally grounded and impactful for 2SLGBTQ+ Lakota youth and their caregivers.

ELIGIBILITY:
Youth Inclusion Criteria:

* Identify as 2SLGBTQ+ (and their identity must be known to their participating caregiver)
* Identify as Indigenous (multiracial youth who are also Indigenous are eligible)
* Youth should be between the ages of 13 and 18 years
* Read and speak English
* Report moderate to high levels of caregiver/family rejection (as evidenced by agreement on items that assess the presence and frequency of specific family rejecting behaviors [includes ambivalent and moderately and highly rejecting caregivers]
* Report an ability and commitment to attending eight sessions at two hours a week over eight weeks with their caregiver

Participating Caregiver Inclusion Criteria:

* Caregivers are broadly defined and may include a biological parent, stepparent, grandparent, aunt/uncle, or other adult who provides care to the Indigenous 2SLGBTQ+ youth
* Must be over the age of 18
* Read and speak English
* Be aware of the SGM identity of their Indigenous 2SLGBTQ+ youth
* report an ability and commitment to attending eight sessions at two hours a week over eight weeks with their teen

Exclusion Criteria:

* We will exclude Indigenous 2SLGBTQ+ youth and caregivers at imminent risk for suicide and/or who are experiencing current psychosis symptoms as determined by results on the safety items screener.

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2026-01-20 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Suicidality (Youth and Caregivers) | Past month at pre-test (enrollment) and post-test (within 1 week of intervention conclusion).
  Participant responses to items from the Suicidal Ideation Attributes Scale to measure suicide and life-threatening behavior in the past month. The 5-item scale includes likert response options ranging from 0 = Never to 10 = Always with higher scores indicating severity of suicidal ideation.
Depression (Youth and Caregivers) | Past 2 weeks at pre-test (enrollment) and post-test (within 1 week of intervention conclusion).
  Participant responses to depressive symptoms in the past two weeks using items from the Patient Health Questionnaire (PHQ-9). The 9-item scale includes likert options ranging from 0 = Not at all to 3 = Nearly every day. Higher scores indicate more depressive symptoms.
Anxiety (Youth and Caregivers) | Past 2 weeks at pre-test (enrollment) and post-test (within 1 week of intervention conclusion).
  Participant responses to items from the Generalized Anxiety Disorder Screener (GAD-7) to measure anxiety symptoms in the past two weeks. The 7-item scale includes likert response options ranging from 0 = not at all to 3 = Nearly every day. Higher scores indicate greater anxiety severity.

SECONDARY OUTCOMES:
Adolescent Dating Violence (Youth) | Past 30 days at pre-test (enrollment) and post-test (within 1 week of intervention conclusion).
  Participant responses to victimization and perpetration experiences in the past 30 days using items from the Adolescent Relationship Harassment and Abuse Scale on the Youth Risk Behavior Survey. The victimization scale is 21 items and the perpetration scale is 24 items. Likert response options range from 0 = 0 times to 3 = More than 10 times. Higher scores indicate greater dating violence.
Alcohol Use (Youth) | Past 30 days pre-test (enrollment) and post-test (within 1 week of intervention conclusion).
  Participant responses to alcohol use items on the Youth Risk Behavior Survey. The 3-item scale assesses alcohol use in the past 30 days. Likert response options for items 1 and 2 range from 0 = 0 days to 6 = all 30 days. Item 3 is an 8 point scale ranging from 0 = I did not drink alcohol in the past 30 days to 8 = 10 or more drinks. Higher scores indicate greater alcohol use.
Drug Use (Youth) | Past 30 days at pre-test (enrollment) and post-test (within 1 week of intervention conclusion).
  Participant responses to items on drug use in the past 30 days from the Youth Risk Behavior Survey. The 8-item scale incudes likert response options ranging from 0 = 0 times to 5 = 40 or more times. Higher scores indicate greater drug use.
School Engagement (Youth) | Collected during the pre-test (enrollment) and post-test (within 1 week of intervention conclusion).
  Participant response to school engagement items from the Hulsey et al., 2018 measure. The 5-item scale includes likert response options ranging from 1= Not at all true of me to 4 = Extremely true of me. Higher scores indicate increased school engagement.
Sexual Risk Taking (Youth) | Past 30 days pre-test (enrollment) and post-test (within 1 week of intervention conclusion).
  Risky Sexual Behavioral Items from the Youth Risk Behavior Survey with participants using a slider to indicate response options ranging from 0 to 100. Higher scores indicate greater sexual risk behavior in the past 30 days.

OTHER OUTCOMES:
(Intermediary Outcome) Caregiver Accepting and Rejecting Behaviors (Youth and Caregivers) | Past 30 days pre-test (enrollment) and post-test (within 1 week of intervention conclusion).
  FAP-Reactions, Advocacy, Feelings/Experiences is a 34 item measure with a 4 point scale for items 1-30 0=Never to 3=Many times. Higher scores indicate more accepting behavior in the past 30 days. A 5 point scale for items 31-32 1=Very Upset to 5=Very Happy with higher scores indicating accepting behavior for item 31 and rejecting behavior for item 32; items 33-34 1=Extremely to 5=Not At All with higher scores indicating accepting behavior for item 33 and rejecting behavior for item 34 in the past 30 days. LGBTQ microaggressions and anti-LGBTQ attitudes (reactions and feelings from microaggressions) subscale is 8 items with a 5 point scale 0=Never to 4=All the time. Higher scores suggest experiencing more interpersonal microaggressions in the past 30 days.
(Intermediary Outcome) Harsh Parenting (Youth and Caregivers) | Collected during the pre-test (enrollment) and post-test (within 1 week of intervention conclusion).
  Items from the Brief Family Relationship Scale to assess family conflict. The 6-item scale includes response options using a continuous slider scale ranging from 1 to 20. Higher scores indicate greater conflict.
(Intermediary Outcome) Connection to Lakota Culture (Youth and Caregivers) | Collected during the pre-test (enrollment) and post-test (within 1 week of intervention conclusion).
  Participant responses to items on the Lakota Cultural Identity Scale. The 7-item scalre includes likert response options ranging from 1 = Not at all to 4 = A lot. Higher scores indicate greater connection to Lakota culture.
(Intermediary Outcome) Connection to Community (Youth and Caregivers) | Collected during the pre-test (enrollment) and post-test (within 1 week of intervention conclusion).
  Participant responses to the Sense of Community Index. The 25-item scale includes likert response options ranging from 1 = Not at all to 4 = Very Important. Higher scores indicate greater sense of community.
(Intermediary Outcome) Ethnic Identity (Youth) | Collected during the pre-test (enrollment) and post-test (within 1 week of intervention conclusion).
  Participant responses to the Multi-group Ethnic Identity Scale. The 12-item scale includes likert response options ranging from 1 = Strongly disagree to 4 = strongly agree. Higher scores indicate greater sense of ethnic identity.
(Intermediary Outcome) Internalized LGBTQ+ phobia (Youth) | Collected during the pre-test (enrollment) and post-test (within 1 week of intervention conclusion).
  Participant responses to the 2017 LGBTQ+ Teen Survey. The 4-item scale includes response options ranging from 1= Strongly Disagree to 4= Strongly agree. Higher scores indicate increased feelings of internalized LGBTQ+ phobia.
(Intermediary Outcome) Lakota Virtues (Youth and Caregivers) | Collected during the pre-test (enrollment) and post-test (within 1 week of intervention conclusion).
  Single item indicator of Lakota virtues that was developed with community input to assess the level of participant agreement with Lakota virtues. The item stem, "My Life Matters" has likert response options that range from 1= strongly disagree to 4= Strongly Agree. Higher scores indicate greater alignment with Lakota virtues.

CONTACTS AND LOCATIONS:
Overall Officials: Katie Edwards, PhD, Principal Investigator — University of Michigan
Locations (2):
- United States (2):
  - Wahwala Iyohlogya/Peaceful Means, Pine Ridge, South Dakota
  - University of Michigan/Rapid City, Rapid City, South Dakota